CLINICAL TRIAL: NCT07180745
Title: Assessment of Efficacy of Empagliflozin Versus Statins in Treatment of Non-Alcoholic Fatty Liver Disease and Non-Alcoholic Steatohepatitis
Brief Title: Empagliflozin Versus Statins in Non-Alcoholic Fatty Liver Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Eman Said Sawan, Lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/01092024
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Non-alcoholic Fatty Liver Disease NAFLD; Non-alcoholic Steatohepatitis NASH
Keywords: Empagliflozin; Statin; Pioglitazone; NAFLD; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Pioglitazone; empagliflozin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Pioglitazone (Active Comparator): 30 mg once daily orally for 3 months
  Interventions: Drug: Pioglitazone (PIO)
- Empagliflozin (Active Comparator): 10 mg once daily orally for 3 months
  Interventions: Drug: Empagliflozin
- Statins (Active Comparator): Once daily orally for 3 months
  Interventions: Drug: Statin (Atorvastatin)
- Empagliflozin plus statins (Active Comparator): Once daily orally for 3 months
  Interventions: Drug: Empagliflozin plus Statin (Atorvastatin)
- Pioglitazone plus Statins (Active Comparator): Once daily orally for 3 months
  Interventions: Drug: Pioglitazone plus Atorvastatin

INTERVENTIONS:
Drug: Pioglitazone (PIO) — 30 mg orally once daily
  Arms: Pioglitazone
Drug: Empagliflozin — 10 mg orally once daily
  Arms: Empagliflozin
Drug: Statin (Atorvastatin) — 20 mg orally once daily
  Arms: Statins
Drug: Empagliflozin plus Statin (Atorvastatin) — Orally once daily of each (10 mg, 20 mg respectively)
  Arms: Empagliflozin plus statins
Drug: Pioglitazone plus Atorvastatin — Orally once daily of each (30mg and 20mg respectively)
  Arms: Pioglitazone plus Statins

SUMMARY:
The goal of this clinical trial is to assess the efficacy of Empagliflozin versus Statins as monotherapy and polytherapy in non-alcoholic fatty liver disease and non-alcoholic Steatohepatitis.

Does drug ABC Empagliflozin versus Statins as monotherapy and polytherapy improve the controlled attenuation parameter (CAP), the liver stiffness measurement (LSM), the proportion of patients with at least one point improvement or one-stage reduction in the histological scores with respect to hepatic steatosis, hepatocellular ballooning, lobular inflammation, and fibrosis after treatment?

What medical problems do participants have when taking Empagliflozin versus Statins as monotherapy and polytherapy?

Participants will:

* Take Empagliflozin alone or Empagliflozin plus statins or Pioglitazone plus Statins or Pioglitazone alone as standard therapy every day for 3 months
* Be directed to complete history taking. FibroScan®, abdominal ultrasound and laboratory tests of ALT, AST, ALP, platelets count, Triglycerides, Cholesterol, LDL, HDL, serum insulin and insulin resistance will be conducted at baseline and after the drug administration for 3 months.
* Keep a diary of recording any side effects they use a rescue inhaler

DETAILED DESCRIPTION:
NAFLD is a growing global health problem linked with metabolic issues like obesity, diabetes, and insulin resistance. It ranges from simple liver fat accumulation to NASH, involving inflammation and liver damage, progressing to fibrosis, cirrhosis, and cancer. Managing NAFLD is tough due to diagnosis challenges and metabolic complications. Lifestyle changes like diet and exercise are key but often hard to sustain. No FDA-approved treatments exist yet, but drugs like Empagliflozin and statins are being studied for their potential to improve insulin sensitivity, reduce liver inflammation, and slow disease progression. This study compares these therapies for NAFLD and NASH.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Obese
* Hyperlipidemic
* Diabetic patients
* Diagnosed with non-alcoholic fatty liver disease and non-alcoholic Steatohepatitis

Exclusion Criteria:

* Pregnant women
* Breast feeding women
* Diabetic patients with ketoacidosis
* Hyperlipidemic patients with cardiovascular dysfunction
* Patients with NAFLD or NASH induced hepatocellular carcinoma
* Hyperlipidemic obese diabetic patients diagnosed with NAFLD or NASH who will refuse to sign the informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The controlled attenuation parameter (CAP). | After 3 months
  The CAP value is expressed in dB/m.
The liver stiffness measurement (LSM) using FibroScan®. | After 3 months
  The LSM value is expressed as kilopascal or kPa.

SECONDARY OUTCOMES:
Fibrosis-4 (FIB-4) index | After 3 months
  FIB-4 is a non-invasive scoring system that can predict significant hepatic fibrosis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Swan, Principal Investigator — Badr University in Cairo, Faculty of Pharmacy
Locations (1):
- Teaching hospital of Beni Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No
Data is available with corresponding author on reasonable request